CLINICAL TRIAL: NCT03537690
Title: A Phase I Study of FID-007 in Patients With Advanced Solid Tumors
Brief Title: FID-007 in Treating Participants With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0C-18-2; NCI-2018-00758 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0C-18-2 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Advanced Malignant Solid Neoplasm; Refractory Malignant Solid Neoplasm
MeSH Terms: interventions — Paclitaxel; Pharmacogenomic Variants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (FID-007) (Experimental): Participants receive FID-007 IV over 60 minutes on days 1, 8 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: PEOX-based Polymer Encapsulated Paclitaxel FID-007; Other: Pharmacokinetic Study

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: PEOX-based Polymer Encapsulated Paclitaxel FID-007 — Given IV
  Other Names: Paclitaxel in Polyethyloxazoline Polymer; FID-007; FID007 (CN); FID 007; Nanoencapsulated Paclitaxel FID-007
Other: Pharmacokinetic Study — Correlative studies
  Other Names: PHARMACOKINETIC; PK Study

SUMMARY:
This phase I trial studies the side effects and best dose of PEOX-based polymer encapsulated paclitaxel FID-007 (FID-007) in treating participants with malignant neoplasms that have spread to other places in the body and do not respond to treatment. FID-007 is a packaged form of the chemotherapy drug paclitaxel, and uses a polyethylozaxoline (PEOX) polymer which may allow the drug to reach deeper into tumors and less into normal cells by being smaller.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of FID-007 and the recommended phase II dose (RP2D).

II. To determine the pharmacokinetics of paclitaxel, (free and total) in patients treated with FID-007.

SECONDARY OBJECTIVES:

I. To characterize the safety and tolerability of FID-007 by assessing toxicities per Common Terminology Criteria for Adverse Events (CTCAE) version (v.)4.3.

II. To obtain a preliminary assessment of anti-tumor activity of FID-007 via objective radiologic tumor response using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

EXPLORATORY OBJECTIVES:

I. To evaluate in a preliminary fashion the serum concentration of total paclitaxel and free paclitaxel, and explore potential associations with serum concentrations, efficacy and toxicity.

OUTLINE: This is a dose escalation study.

Participants receive FID-007 intravenously (IV) over 60 minutes on days 1, 8 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, participants are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histopathologically /cytologically confirmed advanced solid tumor which is refractory to standard therapeutic options, or for which there are no standard therapeutic options, or for whom paclitaxel is an appropriate palliative treatment option (patients for whom paclitaxel or nab-paclitaxel are established treatment options with a proven survival benefit in first line will be excluded)
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status ? 2
* Patient must have recovered from any toxic effects of previous chemotherapy, targeted therapy or radiotherapy as judged by the investigator to ? grade 1
* Previous chemotherapy/radiotherapy/targeted therapy should have been completed at least 4 weeks prior to start of FID-007 administration
* Patients must have an estimated life expectancy of at least 3 months
* Female patients of child bearing potential must have negative serum pregnancy test at screening
* Sexually active women, unless surgically sterile (at least 6 months prior to study drug administration) or postmenopausal for at least 12 consecutive months, must use an effective method of avoiding pregnancy (including oral, transdermal, or implanted contraceptives [any hormonal method in conjunction with a secondary method], intrauterine device, female condom with spermicide, diaphragm with spermicide, absolute sexual abstinence, use of condom with spermicide by sexual partner or sterile [at least 6 months prior to study drug administration] sexual partner) for at least 4 weeks prior to study drug administration, during study and up to 30 days or till next chemotherapy cycle; cessation of birth control after this point should be discussed with a responsible physician; investigator will discuss with patient on the above points and the patient agreement will be documented in the source document; the investigator should ensure that the patient is using an effective method of avoiding pregnancy as per protocol; in case of male patients: either patient partners or patients themselves must use an effective method of avoiding pregnancy for at least 4 weeks prior to study drug administration, during study and up to 30 days or till next chemotherapy cycle
* Patients must agree, as part of the informed consent, to provide blood for pharmacokinetics analysis
* Absolute neutrophil count (ANC) ? 1500/mm^3
* Platelet count ? 100,000/mm^3
* Hemoglobin ? 8 g/dL
* Serum creatinine ? 1.5 X upper limit of normal (ULN) OR calculated clearance ? 50 mL/min/1.73 m^2; if using creatinine clearance, actual body weight should be used for calculating creatinine clearance (e.g., using the Cockcroft-Gault formula); for subjects with a body mass index (BMI) > 30 kg/m^2, lean body weight should be used instead
* Total bilirubin ? 1 X ULN (subjects with Gilbert?s disease can have bilirubin of up to 1.5 X ULN)
* Aspartate aminotransferase (AST) / alanine aminotransferase (ALT) < 3 X ULN
* Patients in the dose escalation phase of the study must have measurable or evaluable disease according to RECIST 1.1 criteria

Exclusion Criteria:

* Patients who have had hypersensitivity to paclitaxel or any of its excipients
* Patients must not have received more than 3 prior lines of cytotoxic chemotherapy for advanced disease; treatment with targeted agents or biologic agents such as antibodies as single agents will not count as a line of cytotoxic chemotherapy
* Patient must not have had prior treatment with paclitaxel or nab-paclitaxel
* Patients must not have serious medical risk factors involving any of the major organ systems, or serious psychiatric disorders, which could compromise the subject's safety or the study data integrity; these include, but are not limited to: history of interstitial lung disease, slowly progressive dyspnea and unproductive cough, sarcoidosis, silicosis, idiopathic pulmonary fibrosis, pulmonary hypersensitivity pneumonitis or multiple allergies
* Patient must not have a history of the following within 6 months prior to cycle 1 day 1: a myocardial infarction, severe/unstable angina pectoris, coronary/peripheral artery bypass graft, New York Heart Association (NYHA) class III-IV heart failure, uncontrolled hypertension, clinically significant cardiac dysrhythmia or electrocardiogram (ECG) abnormality, cerebrovascular accident, transient ischemic attack, or seizure disorder
* Patients who have pre-existing motor or sensory neuropathy of a severity ? grade 1 by CTCAE v4.0 criteria
* Patients who have known active hepatitis B or C
* Patients who have active infection including known human immunodeficiency virus (HIV) infection
* Patients who have concurrent conditions resulting in immune compromise, including chronic treatment with corticosteroids or other immunosuppressive agents
* Patients who are on therapeutic anticoagulation with warfarin; patients on therapeutic doses of with low molecular weight heparins are eligible
* Patients who have ongoing cardiac dysrhythmias, atrial fibrillation, or prolongation of corrected QTc interval to > 480 msec on 2 out of 3 electrocardiograms (EKGs) (if first EKG has QTc < 480, no need to repeat, if first EKG has QTc > 480 repeat twice for a total of 3 EKGs)
* Patients who have known brain metastasis; patients whose central nervous system (CNS) metastases have been treated by surgery or radiotherapy, who are no longer on corticosteroids, and who are neurologically stable are eligible
* Patients for whom paclitaxel (or nab-paclitaxel) is being used in the curative setting, either adjuvant or neoadjuvant, and patients who would receive paclitaxel (or nab-paclitaxel) as first line therapy in a tumor type in which paclitaxel (or nab-paclitaxel) has a proven survival benefit for metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2026-05-25 (Estimated); Study Completion 2027-05-25 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) of PEOX-based polymer encapsulated paclitaxel FID-007 (FID-007) | After first cycle (28 days)
  Will be evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) version (v)4.03 and summarized by dose level, cycle, organ system and type.
Incidence of adverse events | Up to 2 years
  Will be reported using the CTCAE version 4.03.

SECONDARY OUTCOMES:
Clinical anti-tumor response (Complete Response [CR] and Partial Response [PR]) | Up to 2 years
  Will be evaluated using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony El-Khoueiry, MD, Principal Investigator — University of Southern California
Locations (3):
- United States (3):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital, Newport Beach, California